CLINICAL TRIAL: NCT00003032
Title: A Randomized Trial of High-Dose Chemotherapy and Autologous Stem Cell Therapy Versus Standard Therapy in Women With Metastatic Breast Cancer Who Have Responded to Anthracycline or Taxane-Based Induction Chemotherapy
Brief Title: High Dose Chemotherapy Plus Peripheral Stem Cell Transplantation Compared With Standard Therapy in Treating Women With Metastatic or Recurrent Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA16; CAN-NCIC-MA16; CDR0000065634 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Cisplatin; Cyclophosphamide; Mitoxantrone; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: cyclophosphamide
Drug: mitoxantrone hydrochloride
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known whether standard therapy is more effective than high dose chemotherapy for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of high dose chemotherapy plus peripheral stem cell transplantation with that of standard therapy in treating women with metastatic or recurrent breast cancer that has responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival of women with metastatic breast cancer receiving either high dose chemotherapy and autologous peripheral blood stem cell therapy or standard therapy following response to anthracycline or taxane based chemotherapy. II. Evaluate the final response rates between the two treatment arms. III. Compare the two treatment arms with respect to toxic effects. IV. Assess health related quality of life in both groups of patients.

OUTLINE: This is a multicenter, nonblinded, randomized study. Patients are stratified by type of induction chemotherapy, response status, presence of visceral disease, receptor status and tamoxifen therapy (ER negative; ER positive, no prior tamoxifen; ER positive, failed tamoxifen; receptor status unknown). A quality of life questionnaire is given to each patient before and during treatment, then every 3 months thereafter. Patients are assessed following 4 courses of induction chemotherapy. Those achieving complete remission, partial remission, or who have no evaluable disease are randomized to either treatment arm I or arm II. For treatment arm I, stem cells are mobilized by chemotherapy (courses 5 and 6) plus filgrastim (G-CSF) or with G-CSF alone. Following course 6, patients receive daily doses of IV cyclophosphamide, mitoxantrone, and carboplatin on days -6 to -3, followed by stem cell infusion on day 0 and G-CSF from day 5. In arm II, patients receive two further courses of standard induction chemotherapy, followed by maintenance chemotherapy at the discretion of the treating physician. All patients with positive receptor status or unknown receptor status who have not previously failed tamoxifen therapy, receive tamoxifen at the completion of post peripheral stem cell transplant (arm I) or induction chemotherapy (arm II). Following hematologic recovery from high dose chemotherapy patients in arm I with limited disease receive consolidated radiation and may also receive surgical treatment for limited disease. In arm II, patients who completed courses 5 and 6 of induction chemotherapy receive involved field radiation at the physician's discretion. Patients from arm II may also receive surgical treatment following protocol therapy at the physician's discretion. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: This study will accrue approximately 50 patients per year for a total of 192 patients in 3.8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed breast cancer Metastatic disease and/or axillary node or chest wall recurrence following mastectomy diagnosed at least 3 months since prior adjuvant chemotherapy Radiologic scans required No inflammatory carcinoma of the breast without metastases (i.e. T4d M0) No previously untreated inflammatory carcinoma of the breast (T4d) No recurrent breast cancer diagnosed less than 3 months since prior adjuvant chemotherapy No history or evidence of CNS (brain or leptomeningeal) metastases Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 16 to 60 Sex: Female Performance status: ECOG 0-2 Menopausal status: Not specified Life expectancy: Not specified Hematopoietic: Hemoglobin at least 100 g/L Granulocyte count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: AST and/or ALT no greater than 3 times upper limit of normal OR AST and/or ALT no greater than 5 times upper limit of normal, if liver metastases Bilirubin no greater than 1.5 times upper limit of normal Renal: Serum creatinine no greater than 2 times upper limit of normal Cardiovascular: No history of congestive heart failure OR At least 1 year since prior myocardial infarction LVEF at least 45% or normal (ECHO or MUGA are acceptable) Other: No prior or concurrent malignancies allowed, except adequately treated squamous or basal cell carcinoma of the skin or in situ carcinoma of the cervix, or cancer treated more than 5 years ago and presumed cured Not HIV positive No clinical evidence of AIDS Not pregnant or nursing Effective contraception required of fertile patients No major medical illness precluding safe administration of planned treatment or required follow-up

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic response modifier therapy Chemotherapy: No prior chemotherapy for metastatic or recurrent breast cancer Induction chemotherapy required Endocrine therapy: Prior hormonal therapy allowed No concurrent hormonal therapy Radiotherapy: Concurrent radiotherapy allowed for pain control or to solitary bone or soft tissue sites Surgery: Prior oophorectomy allowed See Disease Characteristics

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 224 (Actual)
Dates: Start 1997-04-25 (Actual); Primary Completion 2001-04-12 (Actual); Study Completion 2008-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Crump, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (25):
- Canada (25):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hotel Dieu Hospital - St. Catharines, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - L'Hotel Dieu de Levis, Lévis, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Pavillion de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crump M, Gluck S, Tu D, Stewart D, Levine M, Kirkbride P, Dancey J, O'Reilly S, Shore T, Couban S, Girouard C, Marlin S, Shepherd L, Pritchard KI. Randomized trial of high-dose chemotherapy with autologous peripheral-blood stem-cell support compared with standard-dose chemotherapy in women with metastatic breast cancer: NCIC MA.16. J Clin Oncol. 2008 Jan 1;26(1):37-43. doi: 10.1200/JCO.2007.11.8851. Epub 2007 Nov 19. PMID 18025439
- [Result] Dancey J, Crump M, Gluck S, et al.: Quality of life (QOL) analysis of a randomized trial of high-dose chemotherapy (HDCT) with peripheral stem cell transplant (PSCT) versus standard chemotherapy (SCT) in women with metastatic breast cancer (MBC): National Cancer Institute of Canada Clinical Trials Group study (NCIC CTG) MA-16 . [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-3010, 749, 2003.